CLINICAL TRIAL: NCT03902756
Title: Comparison Between Two Endotracheal Tube Cuff Inflation Methods; Flow Volume Loop Guided vs. Just Seal by Stethoscope Guided in Pediatric Patients
Brief Title: Comparison Between Two Endotracheal Tube Cuff Inflation Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Witchaya Supaopaspan, Principal investigator, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 04-61-24ว
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Endotracheal Cuff Pressure; Flow-Volume Loop Guided; Stethoscope-guided

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flow-Volume loop guided endotracheal cuff inflation (Experimental): Endotracheal cuff will be inflated by Flow-Volume loop guided until getting proper sealing.
  Interventions: Other: Endotracheal cuff inflation
- Stethoscope-guided endotracheal cuff infration (Active Comparator): Endotracheal cuff will be inflated by Stethoscope-guided until getting proper sealing.
  Interventions: Other: Endotracheal cuff inflation

INTERVENTIONS:
Other: Endotracheal cuff inflation — Endotracheal cuff inflation is putting the air in to the endotracheal tube cuff to make the proper sealing.

SUMMARY:
This study is a prospective randomized controlled trial, the primary aim of this study to compare the intracuff pressure which is performed by 2 inflation methods. ( study in pediatric patients 4-12 year old) Group1 : Flow -Volume Loop-guided cuff inflation Group2 : Stethoscope-guided cuff inflation Our hypothesis is Flow-Volume Loop-guided cuff pressure will be lower than Stethoscope-guided cuff pressure.

This study also collect the incidence of common post-extubation respiratory adverse events coughing, hoarseness, stridor, croup as an secondary outcomes.

DETAILED DESCRIPTION:
Historically, pediatric anesthesiologists abstained from using cuff-endotracheal tubes in children younger than 8 year of age because of the anatomical particularises of their airway and thus the increased risk of postintubation tracheal damage especially when Nitrous oxide is used for long procedures. In addition the tube size shoud be half size reduced when cuffed endotracheal tube is used, leading to higher airway resistance and increased risk of tube obstruction.

Recently, the use of Cuffed endotracheal tube has been increasing in children younger than 8 year of age who undergoing general anesthesia. Due to several reasons as follows 1) an increasingly sophisticated understanding of developing laryngeal anatomy 2) vastly improved materials in the manufacture of endotracheal tubes 3) cuffed endotracheal tubes serve several advantages over uncuffed endotracheal tubes including fewer laryngoscopies to replace ill-fitting tubes, less contamination of operating room with anesthetic gases, reliable capnography monitoring, better protection against aspiration, adequate ventilation with a low fresh gas flow which allow using low flow anesthsia, and also they are advantageous for certain operations such as laparoscopic/ airway procedures. 4) data are plentiful supporting the equal safety of using cuffed endotracheal tubes compared with uncuffed tubes in children However, using cuffed endotracheal tubes without being careful of cuff pressure may result in damage to tracheal mucosal wall especially in pediatric patients. The intra-cuff pressure should be monitored and maintained at the level below 25 cm H2O. The intra-cuff pressure more than 30 cmH2O causes obstruction to mucosal blood flow and increasing the risk of airway mucosal injury. Cuff pressure measurement by manometer is a gold standard, nevertheless manometer is not available in every operating room. Almost of anesthetists often use either manual palpation of pilot balloon or stethoscope-guided to inflate endotracheal tube cuff.

In adult studies, they found that endotracheal tube cuff pressure estimated by palpation even with experience personals is often much higher than 25-30 cmH2O. Therefore this inflation technique should be avoided in pediatric patients.

As for, stethoscope-guided endotracheal cuff inflation which pediatric anesthesiologists usually use for children. There were several studies in adult patients, they found the median cuff pressure from this inflation technique was 20 (16-28) cmH2O which is in acceptable tracheal cuff pressure.

In routine practice of general anesthesia rarely have continuous cuff pressure monitoring. When Nitrous Oxide is used for general anesthesia, the intra-cuff pressure can increase with time. Accordingly, it will be better to keep intra-cuff pressure as low as having proper sealing.

A couple studies from adult, compared endotracheal tube cuff inflation techniques between Pressure-Volume(PV) loop guided and stethoscope-guided and the results were intra-cuff pressure from PV loop guided was less than stethoscope guided. Moreover cuff-related complications ( coughing, sorethroat) were less in PV loop group also. It seems PV loop guided can provide least cuff pressure with efficient sealing.

This study would like to compare endotracheal cuff pressure that are performed by 2 techniques between Flow-Volume(FV) loop guided and stethoscope-guided in pediatric patients Intra-cuff pressure will be the primary outcome and we will also collect postoperative respiratory complications such as coughing, stridor, hoarseness as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients are undergoing an operations in Ramathibodi hospital.
* American Society of Anesthesiologists physical status class 1-2
* Endotracheal tube intubation is needed for an operation
* Consent to participate in research project.

Exclusion Criteria:

* Patient who is a predicted difficult intubation
* Patient who has lung disease, airwar abnormalities
* Patient who has pulmonary aspiration risk
* Patient who has a previous sorethroat, hoarseness, respiratory tract infection in last 2 weeks
* Refused to participate in research project

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Intra-cuff pressure | Immediately after cuff inflation
  measuring intra-cuff pressure of endotracheal tube by manometer (cm H2O)

SECONDARY OUTCOMES:
Coughing | 24 hours after extubation
  incidence of coughing
Hoarseness | 24 hours after extubation
  incidence of hoarseness
Stridor | 24 hours after extubation
  incidence of stridor

CONTACTS AND LOCATIONS:
Overall Officials: Witchaya Supaopaspan, medical, Principal Investigator — Mahidol University
Locations (1):
- Ramathibodi Hospital, Bangkok, Ratchathewi, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Orange FA, Andrade RG, Lemos A, Borges PS, Figueiroa JN, Kovatsis PG. Cuffed versus uncuffed endotracheal tubes for general anaesthesia in children aged eight years and under. Cochrane Database Syst Rev. 2017 Nov 17;11(11):CD011954. doi: 10.1002/14651858.CD011954.pub2. PMID 29149469
- [Background] Holzki J, Brown KA, Carroll RG, Cote CJ. The anatomy of the pediatric airway: Has our knowledge changed in 120 years? A review of historic and recent investigations of the anatomy of the pediatric larynx. Paediatr Anaesth. 2018 Jan;28(1):13-22. doi: 10.1111/pan.13281. Epub 2017 Nov 17. PMID 29148119
- [Background] Litman RS, Weissend EE, Shibata D, Westesson PL. Developmental changes of laryngeal dimensions in unparalyzed, sedated children. Anesthesiology. 2003 Jan;98(1):41-5. doi: 10.1097/00000542-200301000-00010. PMID 12502977
- [Background] Tobias JD. Pediatric airway anatomy may not be what we thought: implications for clinical practice and the use of cuffed endotracheal tubes. Paediatr Anaesth. 2015 Jan;25(1):9-19. doi: 10.1111/pan.12528. Epub 2014 Sep 20. PMID 25243638
- [Background] Dalal PG, Murray D, Feng A, Molter D, McAllister J. Upper airway dimensions in children using rigid video-bronchoscopy and a computer software: description of a measurement technique. Paediatr Anaesth. 2008 Jul;18(7):645-53. doi: 10.1111/j.1460-9592.2008.02533.x. Epub 2008 May 8. PMID 18482248
- [Background] Dalal PG, Murray D, Messner AH, Feng A, McAllister J, Molter D. Pediatric laryngeal dimensions: an age-based analysis. Anesth Analg. 2009 May;108(5):1475-9. doi: 10.1213/ane.0b013e31819d1d99. PMID 19372324
- [Background] Litman RS, Maxwell LG. Cuffed versus uncuffed endotracheal tubes in pediatric anesthesia: the debate should finally end. Anesthesiology. 2013 Mar;118(3):500-1. doi: 10.1097/ALN.0b013e318282cc8f. No abstract available. PMID 23314108
- [Background] Weiss M, Dullenkopf A, Fischer JE, Keller C, Gerber AC; European Paediatric Endotracheal Intubation Study Group. Prospective randomized controlled multi-centre trial of cuffed or uncuffed endotracheal tubes in small children. Br J Anaesth. 2009 Dec;103(6):867-73. doi: 10.1093/bja/aep290. Epub 2009 Nov 3. PMID 19887533
- [Background] Shi F, Xiao Y, Xiong W, Zhou Q, Huang X. Cuffed versus uncuffed endotracheal tubes in children: a meta-analysis. J Anesth. 2016 Feb;30(1):3-11. doi: 10.1007/s00540-015-2062-4. Epub 2015 Aug 22. PMID 26296534
- [Background] Gopalareddy V, He Z, Soundar S, Bolling L, Shah M, Penfil S, McCloskey JJ, Mehta DI. Assessment of the prevalence of microaspiration by gastric pepsin in the airway of ventilated children. Acta Paediatr. 2008 Jan;97(1):55-60. doi: 10.1111/j.1651-2227.2007.00578.x. Epub 2007 Dec 10. PMID 18076720
- [Background] Apfelbaum JL, Caplan RA, Barker SJ, Connis RT, Cowles C, Ehrenwerth J, Nickinovich DG, Pritchard D, Roberson DW, Caplan RA, Barker SJ, Connis RT, Cowles C, de Richemond AL, Ehrenwerth J, Nickinovich DG, Pritchard D, Roberson DW, Wolf GL; American Society of Anesthesiologists Task Force on Operating Room Fires. Practice advisory for the prevention and management of operating room fires: an updated report by the American Society of Anesthesiologists Task Force on Operating Room Fires. Anesthesiology. 2013 Feb;118(2):271-90. doi: 10.1097/ALN.0b013e31827773d2. No abstract available. PMID 23287706
- [Background] Black AE, Hatch DJ, Nauth-Misir N. Complications of nasotracheal intubation in neonates, infants and children: a review of 4 years' experience in a children's hospital. Br J Anaesth. 1990 Oct;65(4):461-7. doi: 10.1093/bja/65.4.461. PMID 2248814
- [Background] Dullenkopf A, Schmitz A, Gerber AC, Weiss M. Tracheal sealing characteristics of pediatric cuffed tracheal tubes. Paediatr Anaesth. 2004 Oct;14(10):825-30. doi: 10.1111/j.1460-9592.2004.01316.x. PMID 15385010
- [Background] Seegobin RD, van Hasselt GL. Endotracheal cuff pressure and tracheal mucosal blood flow: endoscopic study of effects of four large volume cuffs. Br Med J (Clin Res Ed). 1984 Mar 31;288(6422):965-8. doi: 10.1136/bmj.288.6422.965. PMID 6423162
- [Background] Liu J, Zhang X, Gong W, Li S, Wang F, Fu S, Zhang M, Hang Y. Correlations between controlled endotracheal tube cuff pressure and postprocedural complications: a multicenter study. Anesth Analg. 2010 Nov;111(5):1133-7. doi: 10.1213/ANE.0b013e3181f2ecc7. Epub 2010 Aug 24. PMID 20736432
- [Background] Borhazowal R, Harde M, Bhadade R, Dave S, Aswar SG. Comparison between Two Endotracheal Tube Cuff Inflation Methods; Just-Seal Vs. Stethoscope-Guided. J Clin Diagn Res. 2017 Jun;11(6):UC01-UC03. doi: 10.7860/JCDR/2017/26301.10017. Epub 2017 Jun 1. PMID 28764268
- [Background] Hoffman RJ, Parwani V, Hahn IH. Experienced emergency medicine physicians cannot safely inflate or estimate endotracheal tube cuff pressure using standard techniques. Am J Emerg Med. 2006 Mar;24(2):139-43. doi: 10.1016/j.ajem.2005.07.016. PMID 16490640
- [Background] Felten ML, Schmautz E, Delaporte-Cerceau S, Orliaguet GA, Carli PA. Endotracheal tube cuff pressure is unpredictable in children. Anesth Analg. 2003 Dec;97(6):1612-1616. doi: 10.1213/01.ANE.0000087882.04234.11. PMID 14633529
- [Background] Kumar RD, Hirsch NP. Clinical evaluation of stethoscope-guided inflation of tracheal tube cuffs. Anaesthesia. 2011 Nov;66(11):1012-6. doi: 10.1111/j.1365-2044.2011.06853.x. Epub 2011 Aug 18. PMID 21851343
- [Background] Almarakbi WA, Kaki AM. Tracheal tube cuff inflation guided by pressure volume loop closure associated with lower postoperative cuff-related complications: Prospective, randomized clinical trial. Saudi J Anaesth. 2014 Jul;8(3):328-34. doi: 10.4103/1658-354X.136422. PMID 25191181
- [Background] Duracher C, Schmautz E, Martinon C, Faivre J, Carli P, Orliaguet G. Evaluation of cuffed tracheal tube size predicted using the Khine formula in children. Paediatr Anaesth. 2008 Feb;18(2):113-8. doi: 10.1111/j.1460-9592.2007.02382.x. PMID 18184241
- [Background] Khine HH, Corddry DH, Kettrick RG, Martin TM, McCloskey JJ, Rose JB, Theroux MC, Zagnoev M. Comparison of cuffed and uncuffed endotracheal tubes in young children during general anesthesia. Anesthesiology. 1997 Mar;86(3):627-31; discussion 27A. doi: 10.1097/00000542-199703000-00015. PMID 9066329
- [Derived] Supaopaspan W, Phongdara S, Vijitpavan A. Endotracheal Tube Cuff Inflation Methods in School-Age Children: Flow-Volume Loop-Guided Versus Stethoscope-Guided. Respir Care. 2025 Feb;70(2):176-183. doi: 10.1089/respcare.12076. PMID 39964846